CLINICAL TRIAL: NCT02035592
Title: The Effects of Blueberry Anthocyanins on Insulin Resistance and Vascular, Lung and Cognitive Function in a Population With Metabolic Syndrome.
Brief Title: The Health Effects of Blueberry Anthocyanins in Metabolic Syndrome (the CIRCLES-study)
Acronym: CIRCLES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of East Anglia (Other)
Collaborators: Harvard School of Public Health (HSPH) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: R21478-C
Record Dates: First submitted 2014-01-10; First posted 2014-01-14 (Estimated); Last update posted 2017-09-29 (Actual); Status verified 2017-01

CONDITIONS: Insulin Resistance; Metabolic Syndrome X
MeSH Terms: conditions — Insulin Resistance; Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Full dose blueberry (Active Comparator): 26g of freeze dried blueberry powder; equivalent to 2 portions of fresh blueberries per day.
  Frequency: 26g per day.
  Total duration: 6-month.
  Interventions: Other: Full dose blueberry
- Half dose blueberry (Active Comparator): 26g of freeze dried powder; containing 13g of freeze dried blueberry powder and 13g of placebo comparator material; equivalent to 1 portion of fresh blueberries per day.
  Frequency: 26g per day.
  Total duration: 6-month.
  Interventions: Other: Half dose blueberry
- Control (Placebo Comparator): Matched control powder; matched for appearance, taste and sugar content.
  Frequency: 26g per day.
  Total duration: 6-month.
  Interventions: Other: Control

INTERVENTIONS:
Other: Full dose blueberry — Full dose: 26g of freeze dried blueberry powder to be incorporated into the habitual diet.
  Dietary restrictions will be observed (i.e. avoidance of blueberry, and restricted intake of anthocyanin rich foods) for 21 days prior to the first assessment visit and throughout the study.
  Arms: Full dose blueberry
Other: Half dose blueberry — Half dose: 26g of freeze dried powder (containing 13g of freeze dried blueberry powder and 13g of placebo comparator material) to be incorporated into the habitual diet.
  Dietary restrictions will be observed (i.e. avoidance of blueberry, and restricted intake of anthocyanin rich foods) for 21 days prior to the first assessment visit and throughout the study.
  Arms: Half dose blueberry
Other: Control — Control: 26g of placebo comparator material to be incorporated into the habitual diet.
  Dietary restrictions will be observed (i.e. avoidance of blueberry, and restricted intake of anthocyanin rich foods) for 21 days prior to the first assessment visit and throughout the study.
  Arms: Control

SUMMARY:
The purpose of this study is to determine the dose-dependent impact of 6 month freeze-dried blueberry powder intake on insulin sensitivity and resistance, cardiovascular disease risk factors, and lung and cognitive function in overweight and obese participants with metabolic syndrome. We will also examine acute post-prandial effects of blueberry intake (at baseline and at 6-months).

ELIGIBILITY:
Inclusion Criteria:

* Men and postmenopausal women (≥ 1 year since last menstruation)
* 50 to 75 years old
* BMI of ≥ 25 kg/m2
* 3 characteristics of metabolic syndrome i.e: Waist circumference ≥ 102 cm for men, ≥ 88 cm for women; Triglycerides ≥ 1.7 mmol/L (or drug treatment for elevated triglycerides); HDL-cholesterol < 1.0 mmol/L for men, < 1.3 mmol/L for women (or drug treatment for low HDL-cholesterol); Blood pressure ≥ 130 mm Hg systolic and/or ≥ 85 mm Hg diastolic blood pressure; Fasting blood glucose ≥ 5.56 mmol/L
* Successful biochemical, haematological and urinalysis assessment at screening

Exclusion Criteria:

* Current smokers, or ex-smokers ceasing < 6 months ago
* Existing or significant past medical history of vascular disease or medical conditions likely to affect the study measures
* Fructose intolerance or known allergies to the intervention treatments
* On therapeutic diets or having experienced substantial weight loss within 3 months of screening
* Taking flavonoid containing supplements (and unwilling to cease intake during, and 1 month preceding the trial)
* Planning on altering consumption of vitamin supplements / fish oil capsules during the course of the study.
* Prescribed hypoglycaemic, vasodilators or HRT medication.
* Unsatisfactory biochemical, haematological or urinary assessment at screening, or measures considered to be counter indicative for the study
* < 3 characteristics of the metabolic syndrome.

NB: REC approved NoSA granted to include those on anti-hypertensives (29JUL2014)

Ages: 50 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2014-01; Primary Completion 2016-11-07 (Actual); Study Completion 2016-11-07 (Actual)

PRIMARY OUTCOMES:
Insulin resistance | Chronic (0 to 6 month)
  Assessed, in the fasted state, via HOMA-IR calculation in all participants; indirect assessment.

SECONDARY OUTCOMES:
Insulin resistance | Chronic (0 to 6 month)
  Assessed in a sub-group via hyperinsulinemic euglycaemic clamp.
Blood pressure and blood vessel regulation | Chronic (0 to 6 month)
  Measurements taken of arterial stiffness, endothelial function and blood pressure.
Lung function | Chronic (0 to 6 month)
  Assessed via standard spirometry techniques and biological assessment of exhaled samples.
Cognitive function | Chronic (0 to 6 month)
  Assessed via a validated cognitive test battery.
Liver fat and blood flow assessment | Chronic (0 to 6 month)
  Assessment via 3T MRI in a sub-group of participants.
Bio-availability | Chronic (0 to 6 month)
  Flavonoid and metabolite levels will be assessed in blood and 24 hour urine samples.
Metabolite phenotype effects | Chronic (0 to 6 month)
  The gut microbiome will be assessed from faecal sample collection and the impact on metabolism and of genotype, will be assessed via a targeted approach.
Acute +24 hour effect of single (26g) intervention intake, given with high fat challenge | Chronic (0 to 6 month)
  Insulin resistance, lipaemia, vascular, cognitive and lung function measured pre- and post-intervention in combination with a high fat challenge in a sub-group of participants. Urine samples and blood samples (over a 24 hour period) will be taken for biomarker analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Aedin Cassidy, PhD, Principal Investigator — University of East Anglia
Locations (4):
- Harvard School of Public Health, Boston, Massachusetts, United States
- United Kingdom (3):
  - Addenbrooke's hospital, Cambridge, Cambridgeshire
  - Norwich Medical School University of East Anglia, Norwich, Norfolk
  - Norfolk and Norwich University Hospital, Norwich, Norfolk

REFERENCES:
- [Derived] Curtis PJ, van der Velpen V, Berends L, Jennings A, Haag L, Minihane AM, Chandra P, Kay CD, Rimm EB, Cassidy A. Chronic and postprandial effect of blueberries on cognitive function, alertness, and mood in participants with metabolic syndrome - results from a six-month, double-blind, randomized controlled trial. Am J Clin Nutr. 2024 Mar;119(3):658-668. doi: 10.1016/j.ajcnut.2023.12.006. Epub 2024 Feb 6. PMID 38432713
- [Derived] Curtis PJ, Berends L, van der Velpen V, Jennings A, Haag L, Chandra P, Kay CD, Rimm EB, Cassidy A. Blueberry anthocyanin intake attenuates the postprandial cardiometabolic effect of an energy-dense food challenge: Results from a double blind, randomized controlled trial in metabolic syndrome participants. Clin Nutr. 2022 Jan;41(1):165-176. doi: 10.1016/j.clnu.2021.11.030. Epub 2021 Nov 27. PMID 34883305
- [Derived] Curtis PJ, van der Velpen V, Berends L, Jennings A, Feelisch M, Umpleby AM, Evans M, Fernandez BO, Meiss MS, Minnion M, Potter J, Minihane AM, Kay CD, Rimm EB, Cassidy A. Blueberries improve biomarkers of cardiometabolic function in participants with metabolic syndrome-results from a 6-month, double-blind, randomized controlled trial. Am J Clin Nutr. 2019 Jun 1;109(6):1535-1545. doi: 10.1093/ajcn/nqy380. PMID 31136659